CLINICAL TRIAL: NCT04402853
Title: SARS Cov-2 in Conjunctival Secretions in an Italian Lombardia Cohort of Patients
Brief Title: SARS Cov-2 in Conjunctival Secretion in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Simone Donati, Associate Professor, Università degli Studi dell'Insubria
Other Study IDs: 72/2020
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Sars-CoV2; Tear
Keywords: COVID 19; EYE; Tears
MeSH Terms: conditions — Lacerations; COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID 19 Patients: hospitalized patients with COVID 19
  Interventions: Diagnostic Test: Tears swab

INTERVENTIONS:
Diagnostic Test: Tears swab — rtPCR on tears swabs samples

SUMMARY:
Observational study to evaluate the presence of SARS COV-2 in tears collected in COVID-19 patients in Lombardia region, northern Italy, and to correlate virus presence to concomitant systemic clinical conditions.

DETAILED DESCRIPTION:
Since February 2020, Coronavirurus Disease 2019 associated to a severe acute respiratory syndrome started in China and rapidly spread all over the world and in particular in northern Italy. There are many reasons to justify this rapid diffusion in Italian Lombardia region as the high population density with more possibilities of interpersonal contact, high prevalence of respiratory pathologies, in particular in elderly people, due to pollution, high number of contacts with Chinese population for travelling and business reasons, and at last the non-windy temperate climate conditions, that increases the persistence of virus in the environment.

At now, more than eighty thousand citizens from Lombardia Region have been officially affected by the disease with a high death toll, also considering that actual numbers are certainly much underestimated.

The aim of the present study was to evaluate the prevalence of SARS COV-2 virus in tears collected from COVID-19 patients by rtPCR analysis directed to target sites of viral RNA, and to correlate virus presence to concomitant systemic clinical conditions

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized COVID 19 patients

Exclusion Criteria:

* Patients with respiratory support that interferes with tears sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with a confirmed diagnosis of COVID 19 pneumonia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Virus presence in COVID 19 patients tears | 1 day
  prevalence of SARS CoV 2 virus on tears

SECONDARY OUTCOMES:
Concordance to Naso-Pharingeal Swab | 1 day
  Evaluation of concordance with Naso-Pharingeal testing

CONTACTS AND LOCATIONS:
Overall Officials: Simone Donati, Professor, Principal Investigator — University of Insubria, Varese
Locations (1):
- ASST Sette Laghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The study will be published

REFERENCES:
- [Background] Wu P, Duan F, Luo C, Liu Q, Qu X, Liang L, Wu K. Characteristics of Ocular Findings of Patients With Coronavirus Disease 2019 (COVID-19) in Hubei Province, China. JAMA Ophthalmol. 2020 May 1;138(5):575-578. doi: 10.1001/jamaophthalmol.2020.1291. PMID 32232433
- [Result] Hong N, Yu W, Xia J, Shen Y, Yap M, Han W. Evaluation of ocular symptoms and tropism of SARS-CoV-2 in patients confirmed with COVID-19. Acta Ophthalmol. 2020 Aug;98(5):e649-e655. doi: 10.1111/aos.14445. Epub 2020 Apr 26. PMID 32336042
- See also: tears and infection — https://www.healio.com/ophthalmology/cornea-external-disease/news/online/%7Bb388d413-6068-4ed7-8a29-f979d33ef1a0%7D/covid-19-possibly-identified-in-tears-conjunctival-secretions